CLINICAL TRIAL: NCT07223411
Title: Dose-response Analysis of Nivolumab/Relatlimab in the Fixed-dosed Combination 'Opdualag' vs. Cemiplimab/Fianlimab in Relation to the Immunological Response in Tumor and Peripheral Blood for Participants With Unresectable or Metastatic Melanoma: A Corollary Study of HCC 24-056 (NCT06246916)
Brief Title: Opdualag vs. Cemiplimab/Fianlimab in Relation to the Immunological Response in Tumor and Peripheral Blood in Unresectable or Metastatic Melanoma
Status: Recruiting | Type: Observational
Sponsor: John Kirkwood (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, John Kirkwood, Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: HCC 25-009
Record Dates: First submitted 2025-10-30; First posted 2025-10-31 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Melanoma
Keywords: immune checkpoint inhibitor; immunological response
MeSH Terms: interventions — cemiplimab; relatlimab; Nivolumab; Opdualag

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- fianlimab + cemiplimab: Patients who received fianlimab + cemiplimab treatment under protocol NCT06246916.
  Interventions: Drug: Fianlimab + Cemiplimab
- Opdualag (relatlimab + nivolumab): Patients who received Opdualag (relatlimab + nivolumab) under protocol NCT06246916.
  Interventions: Drug: Relatlimab + Nivolumab

INTERVENTIONS:
Drug: Fianlimab + Cemiplimab — Patients treated with Fianlimab 1600 mg + Cemiplimab 350 mg under protocol NCT06246916
  Groups: fianlimab + cemiplimab
Drug: Relatlimab + Nivolumab — Patients treated with Relatlimab 160 mg + Nivolumab 480 mg under protocol NCT06246916
  Other Names: Opdualag
  Groups: Opdualag (relatlimab + nivolumab)

SUMMARY:
This translational study will examine the immune effector responses of patients who received a two-drug combination for first line therapy by examining tumor and peripheral blood of participants with unresectable locally advanced or metastatic melanoma.

DETAILED DESCRIPTION:
Cutaneous melanoma is an aggressive skin cancer which, in the metastatic setting, has a historic 5-year survival rate of <30%. In 2023, about 97,610 new cases of melanoma were estimated to occur in the US, with about 7,990 deaths. GLOBACON reported 324,635 cases of melanoma globally in 2020, which constituted about 1.7% of all cancers and 57,043 melanoma-associated deaths.

The parent trial of this corollary study is a randomized, open-label, multicenter phase 3 study comparing the anti-tumor activity of fixed-dose combination (FDC) of fianlimab + cemiplimab versus the FDC of relatlimab + nivolumab (referred to as Opdualag™) in participants with unresectable or metastatic melanoma (stage III-IV). This corollary study will explore the immunological response of CD8, CD4, and other immune cells in the blood and tumor microenvironment of patients in response to the provided treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Study participants who meet inclusion criteria for the HCC 24-056 study will be eligible for this study.
2. Participants must be willing to provide additional samples beyond what is required of them in HCC 24-056. These include:

   1. 3 additional tumor biopsies
   2. 3 additional blood draws
3. Participants must have biopsiable non-target disease amenable to at least 3 biopsies.
4. Must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Study participants who do not qualify to enroll in the HCC 24-056 study will not be eligible for this study.

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study participants who met inclusion criteria for clinical trial NCT06246916
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2031-11-01 (Estimated)

PRIMARY OUTCOMES:
Single-cell analysis of CD4+ T cells | Up to 39 months
  Single-cell RNAseq analysis of CD8+ T cells and other immune cells in blood and tumor biopsies.

SECONDARY OUTCOMES:
Immunological response of CD4+ T cells | Up to 39 months
  Single-cell analysis of CD4+ T cell (frequency) and other immune cells in blood and tumor biopsies. Analysis of single-cell RNA-seq data to obtain gene module scores for each CD4+ T cell or myeloid cell in whole blood and tumor biopsies will be classified as binary: 1 (co-expressing cytotoxic and exhaustion gene modules) or 0 (no co-expression).
Multiplexed immunofluorescence | Up to 39 months
  Degree of immune infiltration major immune subsets in the tumor microenvironment. The density of immune cells relative to the total number of cells in the tumor tissue will be calculated for each patient.
Multiplexed immunofluorescence | Up to 39 months
  Frequencies of major immune subsets in the tumor microenvironment. The density of immune cells relative to the total number of cells in the tumor tissue will be calculated for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: John M Kirkwood, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No